CLINICAL TRIAL: NCT05000788
Title: A Randomized Controlled Neurophysiological Study of Qigong in Elderly With Depression
Brief Title: Neurophysiological RCT of Qigong in Elderly With Depression
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, Dr Yvonne Han, Associate Professor, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HSEARS20210611001
Record Dates: First submitted 2021-05-26; First posted 2021-08-11 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-02

CONDITIONS: Depression
Keywords: Depression; Qigong; Neurophysiology; Functional Near Infra-red Spectroscopy; fNIRS; Executive Function; Attention
MeSH Terms: conditions — Depression | interventions — Qigong; Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Qigong Group (Experimental)
  Interventions: Behavioral: Qigong
- Exercise Group (Active Comparator)
  Interventions: Behavioral: Exercise

INTERVENTIONS:
Behavioral: Qigong — Eight-Section Brocades Practice: The treatment group will undergo an 8-week Eight-Section Brocades intervention program consists of a total of 16 group training sessions with two 1-hour sessions per week. The treatment group participants will be provided with health qigong exercise in a group format led by qualified qigong instructors. All the health qigong instructors will be trained by a certified Traditional Chinese Medicine (TCM) practitioner with an expertise in health qigong and they are required to pass the certification examination before delivering health qigong intervention at the clinical settings. The Eight-Section Brocades protocol will be used in this study because it is easy to learn by the participants and the clinical effects on psychosocial health were evidenced in previous RCTs. A complete cycle of the Eight-Section Brocades took 12 minutes for completion, which consists of eight sequential and simple forms of movements.
  Other Names: Baduanjin
  Arms: Qigong Group
Behavioral: Exercise — Exercise Program: Participants in the control group will attend a physical exercise program for 8 weeks (1-hour sessions, 2 times a week). The exercise program will incorporate aerobic fitness, strength training, body weight workouts, balance training, flexibility and stretching into the training plan. The exercise program is provided in a group format, which will be led by qualified physical trainer.
  Arms: Exercise Group

SUMMARY:
Summary of Project:

Elderly depression is a common mood disorder and the individuals will have persistent low mood and self-absorption that adversely affect their quality of life. Cognitive deficits including attention and executive function are commonly seen in elderly with depression. Qigong, a mind-body practice, is found to have an anti-depressive effect and improve cognitive functions. Yet, the underlying mechanism is still elusive. Hence, the present study aims to conduct a randomized controlled trial to investigate how the practice of Eight-Section Brocades, a type of qigong, affects the function of the central nervous system in elderly with depression, as measured by fNIRS. A total of 60 elderly (based on power analysis 80% (β= 0.20) chance (α = 0.05, two-tailed)), aged 65 or above, with depressive mood as indicated by the Geriatric Depression Scale (GDS) will be recruited and randomly assigned to the treatment (eight-section brocades) and control (exercise) groups. We anticipate that this ancient Chinese mind-body based practice will result in (1) decreased depressive moods and improved cognitive functions, and (2) acute changes in the functional brain activation patterns in the PFC in elderly with depression. The results of this study will shed light on the neurophysiological underpinnings of the therapeutic effects associated with qigong, which will be invaluable for designing intervention for elderly with depression.

ELIGIBILITY:
Inclusion Criteria:

* Elderly aged 65 years or above with depressive symptoms as indicated by the Geriatric Depression Scale (GDS).

Exclusion Criteria:

* Current positive history of head injury, seizure, stroke, other CNS diseases, other comorbid psychiatric illness, or reports of strong suicidal ideation.

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-08-09 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Change in cognitive function as assessed by Attention Network Test | Changes in time points: Baseline, at the end of the 8 weeks, 1 months after treatment
  To evaluate the therapeutic effects of qigong on cognitive functions, we assess a range of cognitive functions including attention, inhibition, and executive function:
  Attention Network Test (ANT). The ANT is a variation from the Flanker test which assesses the efficiency of an individual's subsystems of attention (i.e. alerting, orienting, executive attention). The participants' task is to identify the direction of the central arrow by looking towards the corresponding direction, where either an upward or downward arrow will be presented. The difference of performance between the congruent and incongruent conditions represents inhibitory control ability. Neutral trials will also be presented for measuring simple attention.
Change in cognitive function as assessed by verbal fluency task (VFT) | Changes in time points: Baseline, at the end of the 8 weeks, 1 months after treatment
  Verbal fluency task (VFT). Executive functions are measured using the VFT. The experimental design of this task is adapted from previous fNIRS studies of verbal fluency where task blocks were interleaved with control blocks. Participants are required to generate exemplars of two semantic categories (i.e., animal and means of transportation) as many as possible, each for one minute, during the task blocks. This experimental task will begin with a 30-second phrase repetition period as a control, followed immediately by a 60-second task period (i.e, animal words), a 60-second control period, another 60-second task period (i.e., transportation words), and ended with another 60-second control period. The total measurement period is 270 seconds. The total number of correct and unique responses will be computed to reflect their fluency ability.
Change in cognitive function as assessed by N-back Task | Changes in time points: Baseline, at the end of the 8 weeks, 1 months after treatment
  N-back Task. The N-back paradigm that assesses the updating of working memory is adapted and modified from previous neurophysiological studies that consists of 0-back (i.e., low working memory load), and 2-back (i.e., high working memory load) conditions. Each condition will be presented two times and the tasks will be performed alternately in blocks, separated by a 25-35 seconds rest block during which the participants will be instructed to relax and sit still. The order of the two task blocks will be randomized across participants to avoid order effects, and no condition will be repeated consecutively. Each target (a digit) is presented for 500 milliseconds, followed by an interstimulus interval of 1500 milliseconds. Each task block lasts for 45 seconds, and the total duration of the paradigm is 8 minutes. The accuracy rate and RT of this task will be calculated to reflect the capacity of working memory and processing speed.
Change in executive function as assessed by Cambridge Neuropsychological Test Automated Battery (CANTAB®) | Changes in time points: Baseline, at the end of the 8 weeks, 1 months after treatment
  The CANTAB, a computerised battery of neuropsychological tests, assesses behavioral changes in executive functioning. A test battery that assesses cognitive safety (Roiser et al. 2016) would be used in this study to tap into some of the key cognitive domains. This battery includes four neuropsychological tests which are the (a) Reaction Time (RTI; assesses processing speed and psychomotor speed), (b) Paired Associates Learning (PAL; assesses visual memory and new learning), (c) Spatial Working Memory (SWM, a measure of strategy as well as working memory errors; executive function) and (d) Rapid Visual Information Processing (RVP; assess sustained attention). Also, an emotion recognition task (ERT) which measures the ability to identify emotions in facial expressions will be added to the cognitive safety battery. Six basic emotions will be covered. The total accuracy rate as well as the subscores for different emotions will be recorded to indicate basic emotion recognition ability.
Hemodynamic changes as assessed by functional near-infrared spectroscopy (fNIRS) | Changes in time points: Baseline, at the end of the 8 weeks, 1 months after treatment
  fNIRS is a non-invasive neuroimaging procedure used to measure hemodynamic changes, in terms of oxyhemoglobin (HbO), deoxyhemoglobin (HbR) and total hemoglobin (HbT), associated with neuronal activities of the cerebral cortex in response to attending a task within the given period of time. Optical signals will be recorded on a two-wavelength (780 and 850 nm), continuous-wave optical imaging system (NIRSIT; OBELAB Co., Seoul, South Korea). The 48 channels with a 30-mm source-detector separation which cover the entire PFC area will be used in this study. In accordance with the international 10-20 EEG system, the center of the bottom probe row will be placed at the reference point Fpz. Consequently, channel 1 to channel 16 represent the right PFC, channel 17 to channel 32 the medial PFC, and channel 33 to channel 48 the left PFC. In addition, NIRSIT has an embedded gyroscope that enables online removal of motion artifacts.

SECONDARY OUTCOMES:
Change in mood as assessed by Depression Anxiety Stress Scale-21 (DASS-21) | Changes in time points: Baseline, at the end of the 8 weeks, 1 months after treatment
  The participants' depressive, anxiety, and stress symptoms were evaluated using the 21-item Depression Anxiety Stress Scale [34]. The minimum possible raw score for the depression, anxiety, and stress subscales is 0, while the maximum possible raw score is 21 with higher scores indicating a greater degree of depression, anxiety, and stress. Raw scores on the DASS-21 will need to be multiplied by 2 to calculate the final score for severity labels (normal, mild, moderate, severe, and extremely severe).
Change in mood as assessed by Beck Depression Inventory-II (BDI-II) | Changes in time points: Baseline, at the end of the 8 weeks, 1 months after treatment
  Beck Depression Inventory-II (BDI-II). The participants' severity of depression was also measured using the 21-item Chinese version of the Beck Depression Inventory-II, with higher scores indicating a more severe degree of depression. The possible minimum score is 0, while the possible maximum score is 63.
Change in mood as assessed by Personal Well Being Index (PWI) | Changes in time points: Baseline, at the end of the 8 weeks, 1 months after treatment
  Personal Well Being Index (PWI; Lau et al., 2005). This is an 11-item scale ranging from '0' (extremely dissatisfied) to '10' (extremely satisfied) and used to assess subjective well-being of our participants. The PWI score is the mean of the seven life domains. The study conducted by Lau et al. (2005) showed that it was a reliable measure for use in Hong Kong [36]. The coefficient alpha of PWI was 0.80 and the item-total correlations of PWI ranged between 0.33 and 0.69 for Hong Kong Chinese population.

CONTACTS AND LOCATIONS:
Overall Officials: Hector Tsang, PhD, Study Chair — The Hong Kong Polytechnic University
Locations (1):
- Buddhist Ho L.F. Tak Elderly Social Centre, North Point, HK Island, Hong Kong

IPD SHARING:
Plan to Share IPD: No